CLINICAL TRIAL: NCT03745911
Title: Phase II Study of Paclitaxel and TAK-228 in Metastatic Urothelial Carcinoma (UC) and the Impact of PI3K-mTOR Pathway Genomic Alterations
Brief Title: Paclitaxel and TAK-228 in Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associació per a la Recerca Oncologica, Spain (Other)
Collaborators: Takeda (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X31005; 2017-004486-27 (EudraCT Number)
Record Dates: First submitted 2018-01-09; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Paclitaxel; sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel plus TAK-228 (Experimental): * Paclitaxel will be given on days 1, 8, and 15 of each 28 day cycle intravenously (every Monday or first day of business week if holiday), the day before the first TAK-228 dose. It should be given over approximately one hour.
  * TAK-228 will be given orally on Days 2-4, 9-11, 16-18 and 23-25 of each 28-day cycle.
  Interventions: Combination Product: Paclitaxel and TAK-228

INTERVENTIONS:
Combination Product: Paclitaxel and TAK-228 — Treatment with TAK-228 oral (D2, 3 and 4 of each week) and paclitaxel (D1 of each week) on Days 1, 8 and 15 for each 28-days cycle until disease progression or unacceptable toxicity. If paclitaxel is stopped, TAK-228 may be continued

SUMMARY:
Phase II Multicentre, single arm, open label study of Paclitaxel and TAK-228 in metastatic urothelial carcinoma (UC) and the impact of PI3K-mTOR pathway genomic alterations

DETAILED DESCRIPTION:
The PI3K/AKT/mTOR pathway has been shown to be altered in a large percentage of metastatic urothelial carcinoma (UC) tumors. Within this pathway, the PI3 kinase alpha subunit (PIK3CA) is frequently mutated in muscle invasive bladder cancer (MIBC) (15-20%) and PTEN is inactivated in another 30%.

Due to TAK-228's effects on the PI3K/AKT/mTOR pathway in preclinical studies and the frequency of pathway alterations in UC tumors, TAK-228 is a rational therapy for bladder cancer.

This clinical investigation may also reveal how alterations in the PI3K/AKT/mTOR pathway correlate with treatment response. In preclinical bladder cell line models and xenografts done in our lab, synergistic effect has been seen with the combination with paclitaxel.

The primary end-point is objective response rate (ORR) with the goal of increasing the rate from 10% to 26%. Response rates will be measured using RECIST 1.1 criteria. PFS and OS will be measured from the start date of treatment with TAK-228 and paclitaxel. Grade 3, 4 or serious adverse events will be collected and compared to the catalogued events in the phase II trial in breast cancer (NCT01351350). Patient tumors will be analyzed for genetic alterations within the PI3K/AKT/mTOR pathway to determine if alterations within this pathway correlate with response rate, PFS, or OS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older.
2. Patients must have a diagnosis of metastatic or advanced histologically confirmed UC (urothelial cancer). Mixed histologies are allowed.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Female patients who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 effective method of contraception and 1 additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer as mandated by local labeling [e.g., USPI, SmPC, etc,]) after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).

   Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:
   * Agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).
   * Agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug
5. Screening clinical laboratory values as specified below:

   * Bone marrow reserve consistent with: absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL without transfusion within 1 week preceding study drug administration.
   * Hepatic: total bilirubin ≤ 1.5 x upper limit of normal (ULN), transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase-AST/SGOT and alanine aminotransferase/serum glutamic pyruvic transaminase-ALT/SGPT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present);
   * Renal: creatinine clearance ≥50 mL/min based either on Cockroft-Gault estimate or based on urine collection (12 or 24 hour);
   * Metabolic: Glycosylated hemoglobin (HbA1c) <7.0%, fasting serum glucose (≤ 130 mg/dL) and fasting triglycerides ≤ 300 mg/dL.
6. Ability to swallow oral medications.
7. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
8. Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

   * Brain metastases which have been treated.
   * No evidence of disease progression for ≥3 months before the first dose of study drug.
   * No hemorrhage after treatment.
   * Off-treatment with dexamethasone for 4 weeks before administration of the first dose of TAK-228.
   * No ongoing requirement for dexamethasone or anti-epileptic drugs.
9. Patients having received prior systemic chemotherapy treatment for UC, with no limit for number of prior systemic chemotherapeutic or investigational treatment regimens. Specifically, subjects must meet one or more of the following criteria:

   • Progression after treatment with a regimen that includes a platinum salt (e.g. - carboplatin or cisplatin) for Stage IV disease.

   OR

   • Disease recurrence within one years from the date of last dose of chemotherapy or surgery until day the informed consent is signed) after neoadjuvant or adjuvant treatment with a regimen that includes a platinum salt.
10. Measurable disease, as defined by RECIST v.1.1. If all sites of measurable disease have been irradiated, one site must have demonstrated growth after irradiation.
11. Normal (or within 5% of lower limit) left ventricular ejection fraction

Exclusion Criteria:

1. Prior treatment with paclitaxel for UC (in any setting - neoadjuvant, adjuvant or for metastatic disease). Patients treated with prior docetaxel are eligible.
2. Previous treatment with PI3K, AKT, dual PI3K/mTOR inhibitors, TORC1/2 inhibitors or TORC1 inhibitors.
3. Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of TAK-228. In addition, patients with enteric stomata are also excluded.
4. Poorly controlled diabetes mellitus defined as HbA1c > 7%; subjects with a history of transient glucose intolerance due to corticosteroid administration are allowed in this study if all other inclusion/exclusion criteria are met.
5. Presence of central nervous system metastasis, except for those matching requirements detailed per inclusion criterion 8.
6. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
7. History of any of the following within the last 6 months prior to study entry:

   * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
   * Ischemic cerebrovascular event, including TIA and artery revascularization procedures
   * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
   * Placement of a pacemaker for control of rhythm
   * New York Heart Association (NYHA) Class III or IV heart failure (See Appendix C)
   * Pulmonary embolism.
8. Significant active cardiovascular or pulmonary disease at the time of study entry, including:

   * Uncontrolled high blood pressure (i.e., systolic blood pressure >180 mm Hg, diastolic blood pressure > 95 mm Hg). Use of anti-hypertensive agents to control hypertension before Cycle 1 Day 1 is allowed.
   * Pulmonary hypertension.
   * Uncontrolled asthma or O2 saturation < 90% by ABG (Arterial Blood Gas) analysis or pulse oximetry on room air.
   * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement.
   * Medically significant (symptomatic) bradycardia.
   * History of arrhythmia requiring an implantable cardiac defibrillator.
   * Baseline prolongation of the rate-corrected QT interval (QTc) (e.g., repeated demonstration of QTc interval > 480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes).
9. History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation), which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia.
10. Controlled atrial fibrillation such as with medication or cardioversion is not excluded.
11. Treatment with systemic corticosteroids (either IV or oral steroids, excluding inhalers or low-dose hormone replacement therapy, i.e., prednisone ≤10mg or its equivalent) within 1 week before administration of the first dose of study drug.
12. Women who are currently pregnant or breast feeding.
13. Receipt of any investigational agent, chemotherapy or radiation therapy within 21 days prior to Study Day 1.
14. Any unresolved non-hematologic toxicity greater than CTCAE grade 1 from previous anti-cancer therapy (other than alopecia).
15. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy
16. Grade 2 or greater peripheral neuropathy
17. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
18. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise the patient's participation in the study.
19. Known human immunodeficiency virus infection
20. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
21. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
22. Patients who are taking proton pump inhibitors (PPIs) within 7 days of the first dose of study drug or who require treatment with PPIs throughout the trial or those who are taking H2 receptor antagonists within 24 hours of the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 34 months
  Objective response rate (ORR), defined as the sum of the complete and partial responses (CR+PR), with the goal of increasing the rate from 10% to 26%. Response rates will be measured using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 34 months
  To assess the safety and evaluate the tolerability of TAK-228 in combination with paclitaxel in patients with metastatic, previously treated transitional cell carcinoma.
Progression-Free Survival (PFS) | 34 months
  Time from the first day of therapy to the first evidence of progression as defined by RECIST, or death from any cause, whichever is first. Patients who die without a reported prior progression will be considered to have progressed on the day of their death. Patients alive and without disease progression will be censored at the time of the last objective tumor assessment. Patients who do not progress and are subsequently lost to follow-up will have their data censored at the day of their last objective tumor assessment.
Overall Survival (OS) | 34 months
  Time from the first day of therapy to the date of death from any cause. If the patient is alive at the end of the follow-up period or is lost to follow-up, OS will be censored on the last date the patient is known to be alive.

OTHER OUTCOMES:
Characterization of PI3K/ AKT/ mTOR pathway mutations | 34 months
  Patient tumors samples will be analyzed for genetic alterations within the PI3K/AKT/mTOR pathway to determine if alterations within this pathway correlate with response rate, in patients with UC
Characterization of PI3K/ AKT/ mTOR pathway mutations | 34 months
  Patient tumors samples will be analyzed for genetic alterations within the PI3K/AKT/mTOR pathway to determine if alterations within this pathway correlate with PFS, in patients with UC
Characterization of PI3K/ AKT/ mTOR pathway mutations | 34 months
  Patient tumors samples will be analyzed for genetic alterations within the PI3K/AKT/mTOR pathway to determine if alterations within this pathway correlate with OS, in patients with UC
To discover biomarkers in the serum or plasma (pre and post treatment) of subjects that may predict response to therapy. | 34 months
  Findings suggest S2481 phosphorylation could be a marker for activity of mTORC2. S2481 has the potential to be a prognostic, predictive, and pharmacodynamic marker:
  • Characterize the phosphorylation of S2481 of mTOR in UC tumor tissue
To discover biomarkers in the serum or plasma (pre and post treatment) of subjects that may predict response to therapy. | 34 months
  Findings suggest S2481 phosphorylation could be a marker for activity of mTORC2. S2481 has the potential to be a prognostic, predictive, and pharmacodynamic marker:
  Evaluate whether basal levels of mTOR S2481 phosphorylation correlate with prognosis and/or are predictive of clinical outcomes of the study patients treated with the combination
To discover biomarkers in the serum or plasma (pre and post treatment) of subjects that may predict response to therapy. | 34 months
  Findings suggest S2481 phosphorylation could be a marker for activity of mTORC2. S2481 has the potential to be a prognostic, predictive, and pharmacodynamic marker:
  Assess for changes in tumoral phospho-S2481 after treatment in the biopsy subset of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Bellmunt, MD/PhD, Principal Investigator — Hospital del Mar; Alejo Rodríguez-Vida, MD/PhD, Principal Investigator — Hospital del Mar
Locations (5):
- Spain (5):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Parc Taulí Hospital Universitario, Sabadell, Barcelona
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iyer G, Al-Ahmadie H, Schultz N, Hanrahan AJ, Ostrovnaya I, Balar AV, Kim PH, Lin O, Weinhold N, Sander C, Zabor EC, Janakiraman M, Garcia-Grossman IR, Heguy A, Viale A, Bochner BH, Reuter VE, Bajorin DF, Milowsky MI, Taylor BS, Solit DB. Prevalence and co-occurrence of actionable genomic alterations in high-grade bladder cancer. J Clin Oncol. 2013 Sep 1;31(25):3133-40. doi: 10.1200/JCO.2012.46.5740. Epub 2013 Jul 29. PMID 23897969
- [Background] Guo Y, Chekaluk Y, Zhang J, Du J, Gray NS, Wu CL, Kwiatkowski DJ. TSC1 involvement in bladder cancer: diverse effects and therapeutic implications. J Pathol. 2013 May;230(1):17-27. doi: 10.1002/path.4176. Epub 2013 Mar 21. PMID 23401075
- [Background] Wagle N, Grabiner BC, Van Allen EM, Hodis E, Jacobus S, Supko JG, Stewart M, Choueiri TK, Gandhi L, Cleary JM, Elfiky AA, Taplin ME, Stack EC, Signoretti S, Loda M, Shapiro GI, Sabatini DM, Lander ES, Gabriel SB, Kantoff PW, Garraway LA, Rosenberg JE. Activating mTOR mutations in a patient with an extraordinary response on a phase I trial of everolimus and pazopanib. Cancer Discov. 2014 May;4(5):546-53. doi: 10.1158/2159-8290.CD-13-0353. Epub 2014 Mar 13. PMID 24625776
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Ortmann CA, Mazhar D. Second-line systemic therapy for metastatic urothelial carcinoma of the bladder. Future Oncol. 2013 Nov;9(11):1637-51. doi: 10.2217/fon.13.139. PMID 24156324
- [Background] Vaughn DJ, Broome CM, Hussain M, Gutheil JC, Markowitz AB. Phase II trial of weekly paclitaxel in patients with previously treated advanced urothelial cancer. J Clin Oncol. 2002 Feb 15;20(4):937-40. doi: 10.1200/JCO.2002.20.4.937. PMID 11844814
- [Background] von der Maase H, Sengelov L, Roberts JT, Ricci S, Dogliotti L, Oliver T, Moore MJ, Zimmermann A, Arning M. Long-term survival results of a randomized trial comparing gemcitabine plus cisplatin, with methotrexate, vinblastine, doxorubicin, plus cisplatin in patients with bladder cancer. J Clin Oncol. 2005 Jul 20;23(21):4602-8. doi: 10.1200/JCO.2005.07.757. PMID 16034041
- [Background] Verdoorn BP, Kessler ER, Flaig TW. Targeted therapy in advanced urothelial carcinoma. Oncology (Williston Park). 2013 Mar;27(3):219-26. PMID 23687793
- [Background] Ching CB, Hansel DE. Expanding therapeutic targets in bladder cancer: the PI3K/Akt/mTOR pathway. Lab Invest. 2010 Oct;90(10):1406-14. doi: 10.1038/labinvest.2010.133. Epub 2010 Jul 26. PMID 20661228
- [Background] Platt FM, Hurst CD, Taylor CF, Gregory WM, Harnden P, Knowles MA. Spectrum of phosphatidylinositol 3-kinase pathway gene alterations in bladder cancer. Clin Cancer Res. 2009 Oct 1;15(19):6008-17. doi: 10.1158/1078-0432.CCR-09-0898. Epub 2009 Sep 29. PMID 19789314
- [Background] Bowles DW, Diamond JR, Lam ET, Weekes CD, Astling DP, Anderson RT, Leong S, Gore L, Varella-Garcia M, Vogler BW, Keysar SB, Freas E, Aisner DL, Ren C, Tan AC, Wilhelm F, Maniar M, Eckhardt SG, Messersmith WA, Jimeno A. Phase I study of oral rigosertib (ON 01910.Na), a dual inhibitor of the PI3K and Plk1 pathways, in adult patients with advanced solid malignancies. Clin Cancer Res. 2014 Mar 15;20(6):1656-65. doi: 10.1158/1078-0432.CCR-13-2506. Epub 2014 Feb 3. PMID 24493827
- [Background] Bowles DW, Ma WW, Senzer N, Brahmer JR, Adjei AA, Davies M, Lazar AJ, Vo A, Peterson S, Walker L, Hausman D, Rudin CM, Jimeno A. A multicenter phase 1 study of PX-866 in combination with docetaxel in patients with advanced solid tumours. Br J Cancer. 2013 Sep 3;109(5):1085-92. doi: 10.1038/bjc.2013.474. Epub 2013 Aug 13. PMID 23942080
- [Background] Gomez-Pinillos A, Ferrari AC. mTOR signaling pathway and mTOR inhibitors in cancer therapy. Hematol Oncol Clin North Am. 2012 Jun;26(3):483-505, vii. doi: 10.1016/j.hoc.2012.02.014. Epub 2012 Mar 31. PMID 22520976
- [Background] Seront E, Rottey S, Sautois B, Kerger J, D'Hondt LA, Verschaeve V, Canon JL, Dopchie C, Vandenbulcke JM, Whenham N, Goeminne JC, Clausse M, Verhoeven D, Glorieux P, Branders S, Dupont P, Schoonjans J, Feron O, Machiels JP. Phase II study of everolimus in patients with locally advanced or metastatic transitional cell carcinoma of the urothelial tract: clinical activity, molecular response, and biomarkers. Ann Oncol. 2012 Oct;23(10):2663-2670. doi: 10.1093/annonc/mds057. Epub 2012 Apr 3. PMID 22473592
- [Background] Milowsky, M.I., Final results of a multicenter, open-label phase II trial of dovitinib (TKI258) in patients with advanced urothelial carcinoma with either mutated or nonmutated FGFR3. 2013, J Clin Oncol 2013; 31(Suppl 6) [abstract: 255].
- [Background] Bajorin DF. Paclitaxel in the treatment of advanced urothelial cancer. Oncology (Williston Park). 2000 Jan;14(1):43-52, 57; discussion 58, 61-2. PMID 10680149
- [Background] Raghavan D. Progress in the chemotherapy of metastatic cancer of the urinary tract. Cancer. 2003 Apr 15;97(8 Suppl):2050-5. doi: 10.1002/cncr.11280. PMID 12673696
- [Background] Rossi JF. Phase I study of atacicept in relapsed/refractory multiple myeloma (MM) and Waldenstrom's macroglobulinemia. Clin Lymphoma Myeloma Leuk. 2011 Feb;11(1):136-8. doi: 10.3816/CLML.2011.n.031. PMID 21454215
- [Background] Chiang GG, Abraham RT. Targeting the mTOR signaling network in cancer. Trends Mol Med. 2007 Oct;13(10):433-42. doi: 10.1016/j.molmed.2007.08.001. Epub 2007 Oct 1. PMID 17905659
- [Background] Sabatini DM. mTOR and cancer: insights into a complex relationship. Nat Rev Cancer. 2006 Sep;6(9):729-34. doi: 10.1038/nrc1974. Epub 2006 Aug 17. PMID 16915295
- [Background] Jessen K, Wang S, Kessler L, et al. INK128 is a potent and selective TORC1/2 inhibitor with broad oral antitumor activity. Mol Cancer Ther. 2009;8(12 Suppl) Abstract B148
- [Background] Kessler L, Wang S, Xin G, Kucharski J, Staunton J, Lan L, et al. INK128, an orally active TORC1/2 kinase inhibitor, shows broad antitumor activity and enhances efficacy of cytotoxic as well as targeted agents. Cancer Res 2010;70(8; Supplement 1 Abstract 4496).
- [Background] Hassan B, Akcakanat A, Takafumi S, Evans K, Adkins F, Meric-Bernstam F. Inhibitor MLN0128 Has Antitumor Efficacy In Cell Lines With Intrinsic And Acquired Rapamycin-Resistance. Academic Surgical Congress 2013(Abstract ASC20130420).
- [Background] Shafer A, Zhou C, Gehrig PA, Boggess JF, Bae-Jump VL. Rapamycin potentiates the effects of paclitaxel in endometrial cancer cells through inhibition of cell proliferation and induction of apoptosis. Int J Cancer. 2010 Mar 1;126(5):1144-54. doi: 10.1002/ijc.24837. PMID 19688827
- [Background] Shu CH, Yang WK, Shih YL, Kuo ML, Huang TS. Cell cycle G2/M arrest and activation of cyclin-dependent kinases associated with low-dose paclitaxel-induced sub-G1 apoptosis. Apoptosis. 1997;2(5):463-70. doi: 10.1023/a:1026422111457. PMID 14646529
- [Background] Mondesire WH, Jian W, Zhang H, Ensor J, Hung MC, Mills GB, Meric-Bernstam F. Targeting mammalian target of rapamycin synergistically enhances chemotherapy-induced cytotoxicity in breast cancer cells. Clin Cancer Res. 2004 Oct 15;10(20):7031-42. doi: 10.1158/1078-0432.CCR-04-0361. PMID 15501983
- [Background] Voss M, Gordon MS, Mita M, Rini B, Makker V, Macarulla T, et al. Phase I study of investigational oral mTORC1/2 inhibitor TAK-228 (formerly MLN0128): expansion phase in patients with renal, endometrial, or bladder cancer. ESMO poster Sept 2015
- [Background] Ghobrial IM, Siegel DS, Vij R, Berdeja JG, Richardson PG, Neuwirth R, Patel CG, Zohren F, Wolf JL. TAK-228 (formerly MLN0128), an investigational oral dual TORC1/2 inhibitor: A phase I dose escalation study in patients with relapsed or refractory multiple myeloma, non-Hodgkin lymphoma, or Waldenstrom's macroglobulinemia. Am J Hematol. 2016 Jun;91(4):400-5. doi: 10.1002/ajh.24300. PMID 26800393
- [Background] TAK-228 Investigator Brochure Edition 10. 22 March 2017
- [Background] PACLITAXEL - paclitaxel injection, solution [package insert]. Princeton, NJ. Sandoz; 2011
- [Derived] Hernandez-Prat A, Rodriguez-Vida A, Juanpere-Rodero N, Arpi O, Menendez S, Soria-Jimenez L, Martinez A, Iarchouk N, Rojo F, Albanell J, Brake R, Rovira A, Bellmunt J. Novel Oral mTORC1/2 Inhibitor TAK-228 Has Synergistic Antitumor Effects When Combined with Paclitaxel or PI3Kalpha Inhibitor TAK-117 in Preclinical Bladder Cancer Models. Mol Cancer Res. 2019 Sep;17(9):1931-1944. doi: 10.1158/1541-7786.MCR-18-0923. Epub 2019 Jun 3. PMID 31160383